CLINICAL TRIAL: NCT05218057
Title: TFL vs Ho:YAG - A Prospective Study to Compare the Effectiveness of Thulium Fiber Laser and Holmium YAG Laser for Ureteroscopic Lithotripsy
Brief Title: to Compare the Effectiveness of Thulium Fiber Laser and Holmium YAG Laser for Ureteroscopic Lithotripsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Chi Fai NG, Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CRE 2021.652
Record Dates: First submitted 2021-12-30; First posted 2022-02-01 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Ureteric Stone
MeSH Terms: conditions — Ureterolithiasis

STUDY DESIGN:
Who Masked: Participant
Masking Description: The urologist performing the surgery could not be blinded due to the nature of the intervention. Patients receiving the treatment and investigators assessing for the outcomes are blinded from the allocated treatment arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Thulium-fibre laser (TFL) (Active Comparator): The laser used in this group for surgical procedure ureteroscopic lithotripsy will be the Olympus SOLTIVETM Premium SuperPulsed laser system with a 365micron laser fibre. The laser pulse setting will be 1J x 10Hz, short pulse duration (adjusted up to 600microseconds).
  Interventions: Procedure: Ureteroscopic lithotripsy
- Holmium: yttrium-aluminum-garnet (Ho: YAG) (Active Comparator): The laser used in this group for surgical procedure ureteroscopic lithotripsy will be the Lumenis VersaPulse® PowerSuiteTM 100W laser system with a 365micron laser fibre. The laser pulse setting will be 1J x 10Hz. Pulse duration is not adjustable in this machine (up to 600microseconds).
  Interventions: Procedure: Ureteroscopic lithotripsy

INTERVENTIONS:
Procedure: Ureteroscopic lithotripsy — Ureteroscopic lithotripsy is one of the surgical procedure options for ureteric stone less than 1.5 cm. While many energy systems has been used for stone fragmentation during ureteroscopy, laser energy is the most commonly used approach for stone fragmentation.

SUMMARY:
This prospective randomized clinical trial aimed to compare the difference in stone ablation rates of TFL and Ho:YAG laser in a clinical setting. Patients are randomized to receive URS with lithotripsy (URSL) either with TFL or Ho:YAG with an allocation ratio of 1:1. Primary outcome is the efficiency of stone ablation in terms of the stone ablation rate

DETAILED DESCRIPTION:
Having the advantages of being minimally invasive and simple, ureteroscopic lithotripsy is one of the treatment options for ureteric stone less than 1.5 cm. While many energy systems has been used for stone fragmentation during ureteroscopy, laser energy is the most commonly used approach for stone fragmentation. Currently, Holmium-YAG laser is the main laser platform being used due to its preciseness and safety. Unfortunately, Holmium-YAG laser system has some intrinsic problems, such as lower energy conversion ratio, excessive heat generation in machines, noise etc. Therefore, newer laser systems are being developed to overcome the problem. Thulium-fiber Laser (TFL) is the latest available laser system in the market with promising results. The advantages of TFL included better energy conversion ratio, less heat energy generation, more portable size, allow the generation of higher laser frequency for better stone dusting etc. Therefore, its uses are increasing popular. However, there are not many studies comparing the efficacy and stone free results of the Holmium-YAG laser and TFL systems in the literature. Therefore, investigators would like to perform a formal study to compare the two systems.

.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18-years-old with informed consent

Exclusion Criteria:

* Patients on anti-coagulation
* Patients with condition that increases the risk of urolithiasis (e.g. cystinuria, hyperparathyroidism, previous intestinal resection)
* Patients with abnormal urinary tract (e.g. ileal conduit, neobladder, ureteric stricture)
* Patients with stones > 15 mm

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2023-09-29 (Actual); Study Completion 2023-10-30 (Actual)

PRIMARY OUTCOMES:
The efficiency of stone ablation | Intraoperation
  Measured by stone ablation rate(pre-operative stone volume/ laser time)

SECONDARY OUTCOMES:
Operation time | Intra-operation
  Duration of operation
Laser time | Intra-operation
  Duration of laser use
Length of hospital stay | The total number of days of hospitalization for this surgical procedure up to day 30 after the procedure
  Total number of days of hospitalization for the surgical procedure
Number of patient with Complications after surgical procedure | 30 days post-operation
  Complications of treatment using Common Terminology Criteria for Adverse Events (CTCAE) v5.0
Stone free rate | 3 months post-operation
  Defined by no detectable stone on post-operative 3-month NCCT
Number of patients require auxiliary procedure after the intervention | 3 months post-operation
  Defined by any additional procedure

CONTACTS AND LOCATIONS:
Overall Officials: Chi Fai NG, MD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- North District Hospital, Sheung Shui, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Tae BS, Balpukov U, Cho SY, Jeong CW. Eleven-year Cumulative Incidence and Estimated Lifetime Prevalence of Urolithiasis in Korea: a National Health Insurance Service-National Sample Cohort Based Study. J Korean Med Sci. 2018 Jan 8;33(2):e13. doi: 10.3346/jkms.2018.33.e13. PMID 29215822
- [Background] Ziemba JB, Matlaga BR. Epidemiology and economics of nephrolithiasis. Investig Clin Urol. 2017 Sep;58(5):299-306. doi: 10.4111/icu.2017.58.5.299. Epub 2017 Aug 10. PMID 28868500
- [Background] Sorokin I, Mamoulakis C, Miyazawa K, Rodgers A, Talati J, Lotan Y. Epidemiology of stone disease across the world. World J Urol. 2017 Sep;35(9):1301-1320. doi: 10.1007/s00345-017-2008-6. Epub 2017 Feb 17. PMID 28213860
- [Background] Elashry OM, Tawfik AM. Preventing stone retropulsion during intracorporeal lithotripsy. Nat Rev Urol. 2012 Dec;9(12):691-8. doi: 10.1038/nrurol.2012.204. Epub 2012 Nov 20. PMID 23165399
- [Background] Li JK, Teoh JY, Ng CF. Updates in endourological management of urolithiasis. Int J Urol. 2019 Feb;26(2):172-183. doi: 10.1111/iju.13885. Epub 2018 Dec 21. PMID 30575154
- [Background] Saussine C, Andonian S, Pacik D, Popiolek M, Celia A, Buchholz N, Sountoulides P, Petrut B, de la Rosette JJMCH. Worldwide Use of Antiretropulsive Techniques: Observations from the Clinical Research Office of the Endourological Society Ureteroscopy Global Study. J Endourol. 2018 Apr;32(4):297-303. doi: 10.1089/end.2017.0629. Epub 2018 Jan 17. PMID 29256629
- [Background] Traxer O, Keller EX. Thulium fiber laser: the new player for kidney stone treatment? A comparison with Holmium:YAG laser. World J Urol. 2020 Aug;38(8):1883-1894. doi: 10.1007/s00345-019-02654-5. Epub 2019 Feb 6. PMID 30729311
- [Background] Fried NM. Recent advances in infrared laser lithotripsy [Invited]. Biomed Opt Express. 2018 Aug 30;9(9):4552-4568. doi: 10.1364/BOE.9.004552. eCollection 2018 Sep 1. PMID 30615704
- [Background] Andreeva V, Vinarov A, Yaroslavsky I, Kovalenko A, Vybornov A, Rapoport L, Enikeev D, Sorokin N, Dymov A, Tsarichenko D, Glybochko P, Fried N, Traxer O, Altshuler G, Gapontsev V. Preclinical comparison of superpulse thulium fiber laser and a holmium:YAG laser for lithotripsy. World J Urol. 2020 Feb;38(2):497-503. doi: 10.1007/s00345-019-02785-9. Epub 2019 May 4. PMID 31055626
- [Background] Martov AG, Ergakov DV, Guseynov M, Andronov AS, Plekhanova OA. Clinical Comparison of Super Pulse Thulium Fiber Laser and High-Power Holmium Laser for Ureteral Stone Management. J Endourol. 2021 Jun;35(6):795-800. doi: 10.1089/end.2020.0581. Epub 2021 Jan 13. PMID 33238763
- [Background] Traxer O, Corrales M. Managing Urolithiasis with Thulium Fiber Laser: Updated Real-Life Results-A Systematic Review. J Clin Med. 2021 Jul 30;10(15):3390. doi: 10.3390/jcm10153390. PMID 34362169